CLINICAL TRIAL: NCT03183440
Title: A Multicenter Clinical Trial To Assess The Efficacy Of Antenatal Maternal Supplementation With GOS/Inulin Prebiotics On Atopic Dermatitis Prevalence In High-Risk One-Year-Old Children.
Brief Title: Efficacy Of Antenatal Maternal Supplementation With GOS/Inulin Prebiotics On Atopic Dermatitis Prevalence In High-Risk One-Year-Old Children
Acronym: PREGRALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC16_0012
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatitis; Prevention; Prebiotics; Pregnancy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREBIOTICS (Experimental): 188 pregnant women
  Interventions: Dietary Supplement: PREBIOTICS
- PLACEBO (Placebo Comparator): 188 pregnant women
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: PREBIOTICS — women will daily take a mixture of Galacto-Oligo-Saccharide/inulin (ratio 9:1) from inclusion to delivery
  Arms: PREBIOTICS
Other: PLACEBO — women will daily take placebo (maltodextrin) from inclusion to delivery
  Arms: PLACEBO

SUMMARY:
Allergies are increasing worldwide affecting 30-40% of the population. Among this, Atopic Dermatitis (AD) is the earliest and the most common manifestation of allergic diseases (prevalence 20%). Recent studies have shown that allergies were associated with a disruption of the gut microbial 'balance' suggesting that the use of nutritional intervention very early in life may restore an optimal pattern of microflora aiming at improving the host's health. So far, most human intervention studies have mainly focused on improving postnatal infant colonization. Our study will test the hypothesis that a maternal antenatal prebiotics (GOS/inulin) supplementation may be superior to placebo for AD prevention in high-risk children.

DETAILED DESCRIPTION:
Study design :

Inclusion visit at 20 weeks of gestation :

* randomization
* start of supplementation (GOS/inulin or placebo)

Phone call at 24 weeks of gestation :

* checking tolerance
* checking observance

  32 weeks of gestation visit :
* replenishment of prebiotics
* collect of AE

Day 1 : assessment of the Transepidermal Waterlos evaluated by a TEWAMETER

Delivery/per partum Visit

At M3 : The national recommendations for the dietary diversification of the child will be transmitted to the patients

At M6 : evaluation of AD prevalence by parents

At M12 : Pediatric dermatology consultation

* clinical exam of child
* the SCORAD
* the POEM questionnaire
* prevalence of AD
* skin prick tests
* FDQLI score
* assessment of the Transepidermal Waterlos evaluated by a TEWAMETER
* prevalence of food allergies

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with an eutocic pregnancy before 20 weeks of gestation
* women with personal history of atopy diagnosed by a healthcare Professional
* Women accepting a complete avoidance of dietary supplements containing prebiotics or probiotics during study supplementation
* women accepting dermato-pediatric follow-up during the first year of life of the new-born (Phone calls at 24 weeks of gestation and 6 months of child and a consultation at 12 months of age)
* non Tobacco user women
* women over 18 years
* women without history of severe gestational diabetes

Exclusion Criteria:

* women not giving up on intake of dietary supplements containing prebiotics or probiotics during study supplementation
* women refusing dermato-pediatric follow-up during the first year of the newborn
* ongoing allergy and/or intolerance to cow's milk proteins
* term >21 weeks of gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
atopic dermatitis prevalence at M12 | at 12 months of age
  prevalence will be evaluated according to UK party working group criteria

SECONDARY OUTCOMES:
atopic dermatitis prevalence at M6 | at 6 months of age
  prevalence will be evaluated by a phone questionnaire (ISAAC questionnaire)
atopic dermatitis severity | at 12 months of age
  evaluated by the SCORAD (Scoring Atopic Dermatitis)
atopic dermatitis severity | at 12 months of age
  evaluated by the POEM (Patient Oriented Eczema Measure)
Quality of life of the child and his/her family | at 12 months of age
  evaluated by the FDQLI score (Family Dermatitis Quality of life Index)
Tolerance of the prebiotics in mothers | from inclusion to delivery
  evaluated by a questionnaire on digestive status (bloating, stomach aches, diarrhea, flatulences,...)
sensitization with the major allergens | at 12 months of age
  skin prick tests
assessment of the Transepidermal Waterlos | at J1 and at 12 months of age
  evaluated by a TEWAMETER(R)
food allergies prevalence at M12 | at 12 months of age
  Prevalence will be evaluated by recording food allergies diagnosed by a physician

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Angers, Angers
  - CHD Vendée, La Roche-sur-Yon
  - CHU Nantes, Nantes
  - University Hospital, Rennes
  - Centre Hospitalo Universitaire, Toulouse
  - University Hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barbarot S, Aubert H, Boivin M, Foureau A, Maruani A, Droitcourt C, Mazereeuw-Hautier J, Faurel-Paul E, Le Thuaut A, Tching-Sin M, Dochez V, Brosseau C, Bodinier M. Evaluation of antenatal prebiotic intake in infants at risk of atopy: the double-blind PREGRALL randomized clinical trial. Br J Dermatol. 2025 Nov 18:ljaf414. doi: 10.1093/bjd/ljaf414. Online ahead of print. PMID 41250898
- [Derived] Cabridain C, Aubert H, Kaeffer B, Badon V, Boivin M, Dochez V, Winer N, Faurel-Paul E, Planche L, Riochet D, Maruani A, Perrotin F, Droitcourt C, Lassel L, Tching-Sin M, Rogers NK, Bodinier M, Barbarot S. Effectiveness of an antenatal maternal supplementation with prebiotics for preventing atopic dermatitis in high-risk children (the PREGRALL study): protocol for a randomised controlled trial. BMJ Open. 2019 Apr 20;9(4):e024974. doi: 10.1136/bmjopen-2018-024974. PMID 31005913